CLINICAL TRIAL: NCT00971633
Title: An Open-Label, Randomized, Single Dose, 3-period Crossover Study to Determine the Bioequivalence of 3 Formulations of Ondansetron in Healthy Young Adult Male and Female Subjects
Brief Title: A Bioequivalence Study of 3 Formulations of Ondansetron in Healthy Adults (0869-095)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0869-095; 2009_656
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Treatment Sequence A-B-C
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)
- 2 (Experimental): Treatment Sequence B-C-A
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)
- 3 (Experimental): Treatment Sequence C-A-B
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)
- 4 (Experimental): Treatment Sequence A-C-B
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)
- 5 (Experimental): Treatment Sequence B-A-C
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)
- 6 (Experimental): Treatment Sequence C-B-A
  Interventions: Drug: Comparator: Treatment A (Zofran, ondansetron); Drug: Comparator: Treatment B (Zofran, ondansetron); Drug: Comparator: Treatment C (Zofran, ondansetron)

INTERVENTIONS:
Drug: Comparator: Treatment A (Zofran, ondansetron) — an over-encapsulated single 8 mg tablet of United Kingdom (U.K.) Zofran taken by mouth (PO)
  Other Names: Zofran, ondansetron
Drug: Comparator: Treatment B (Zofran, ondansetron) — a single 8 mg tablet of Zofran marketed in the U.K., taken PO
  Other Names: Zofran, ondansetron
Drug: Comparator: Treatment C (Zofran, ondansetron) — a single 8 mg tablet of Zofran marketed in the United States (U.S.), taken PO
  Other Names: Zofran, ondansetron

SUMMARY:
This study will assess the bioequivalence of a Merck clinical trial formulation of ondansetron compared to a U.S. and non-U.S. marketed formulation of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* If female, subject is not pregnant or breast-feeding
* Subject is a nonsmoker
* Subject is in good general health

Exclusion Criteria:

* Subject has a history of high blood pressure, asthma, or cardiovascular, liver, neurologic, or kidney disease
* Subject is taking prescription or nonprescription drugs that can not be discontinued during the study
* Subject is a habitual and heavy consumer of caffeine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-11; Primary Completion 2003-12 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- OE U.K. Tablet Then U.K. Tablet Then U.S. Tablet: Over-encapsulated (OE) United Kingdom (U.K.) tablet then U.K. tablet then United States (U.S.) tablet: Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of United Kingdom (U.K.) ZOFRAN (ondansetron) taken orally./Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally./Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally
- U.K. Tablet Then U.S. Tablet Then OE U.K. Tablet: U.K. tablet then U.S. tablet then OE U.K. tablet: Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.K. taken orally /Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally/Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of U.K. ZOFRAN (ondansetron) taken orally.
- U.S. Tablet Then OE U.K. Tablet Then U.K. Tablet: U.S. tablet then OE U.K. tablet then U.K. tablet: Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally/Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of U.K ZOFRAN (ondansetron) taken orally/Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.K. taken orally
- OE U.K. Tablet Then U.S. Tablet Then U.K. Tablet: OE U.K. tablet then U.S. tablet then U.K. tablet: Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of U.K. ZOFRAN (ondansetron) taken orally/Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally/Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.K. taken orally
- U.K. Tablet Then OE U.K. Tablet Then U.S. Tablet: U.K. tablet then OE U.K. tablet then U.S. tablet: Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.K. taken orally/Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of U.K. ZOFRAN (ondansetron) taken orally/Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally
- U.S. Tablet Then U.K. Tablet Then OE U.K. Tablet: U.S. tablet then U.K. tablet then OE U.K. tablet: Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.S. taken orally/Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the U.K. taken orally/Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of U.K. ZOFRAN (ondansetron) taken orally
Period: Period 1
Arm/Group | OE U.K. Tablet Then U.K. Tablet Then U.S. Tablet | U.K. Tablet Then U.S. Tablet Then OE U.K. Tablet | U.S. Tablet Then OE U.K. Tablet Then U.K. Tablet | OE U.K. Tablet Then U.S. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet Then U.S. Tablet | U.S. Tablet Then U.K. Tablet Then OE U.K. Tablet
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | OE U.K. Tablet Then U.K. Tablet Then U.S. Tablet | U.K. Tablet Then U.S. Tablet Then OE U.K. Tablet | U.S. Tablet Then OE U.K. Tablet Then U.K. Tablet | OE U.K. Tablet Then U.S. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet Then U.S. Tablet | U.S. Tablet Then U.K. Tablet Then OE U.K. Tablet
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | OE U.K. Tablet Then U.K. Tablet Then U.S. Tablet | U.K. Tablet Then U.S. Tablet Then OE U.K. Tablet | U.S. Tablet Then OE U.K. Tablet Then U.K. Tablet | OE U.K. Tablet Then U.S. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet Then U.S. Tablet | U.S. Tablet Then U.K. Tablet Then OE U.K. Tablet
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 31.7 [25 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Weight [Mean (Full Range); unit: kilograms] | 78.5 [61.1 to 101.0]
Height [Mean (Full Range); unit: centimeters] | 171.1 [155 to 183]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero to Infinity (AUC) of Ondansetron
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 24 hours post dose
Population: All study participants (N=12)
Measure: Least Squares Mean (Standard Deviation); unit: nM*hr
Groups:
- Treatment OE U.K. Tablet: Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of United Kingdom (U.K.) ZOFRAN (ondansetron) taken orally
- Treatment U.K. Tablet: Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally
- Treatment U.S. Tablet: Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United States (U.S.) taken orally
Arm/Group | Treatment OE U.K. Tablet | Treatment U.K. Tablet | Treatment U.S. Tablet
Number analyzed (Participants) | 12 | 12 | 12
nM*hr | 644 (240) | 712 (233) | 649 (255)
Statistical Analysis 1: Comparison: Treatment OE U.K. Tablet vs Treatment U.K. Tablet; Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of United Kingdom (U.K.) ZOFRAN (ondansetron) taken orally Treatment U.K. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally; Test type: Non-Inferiority or Equivalence — Study Secondary Hypothesis: A single dose of U.K. ZOFRAN (ondansetron) 8-mg table over-encapsulated is bioequivalent to a single dose of the U.K. ZOFRAN (ondansetron) 8-mg tablet. That is, the true geometric mean ratios (U.K. ZOFRAN tablet over-encapsulated/U.K. ZOFRAN tablet) of the area under the plasma concentration vs. time curve (AUC) from zero to infinity and maximum plasma concentration (Cmax) for ondansetron each lie within the interval 0.80 to 1.25; Geometric Mean Ratio = 0.904, 95% CI 2-sided [0.796 to 1.028] — Geometric Mean Ratio (Treatment OE U.K. tablet / Treatment U.K. tablet)
Statistical Analysis 2: Comparison: Treatment OE U.K. Tablet vs Treatment U.S. Tablet; Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of United Kingdom (U.K.) ZOFRAN (ondansetron) taken orally Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United States (U.S.) taken orally; Test type: Non-Inferiority or Equivalence — Study Primary Hypothesis: A single dose of the U.K. ZOFRAN (ondansetron) 8-mg tablet over-encapsulated is bioequivalent to a single dose of the U.S. ZOFRAN (ondansetron) 8-mg tablet. That is, the true geometric mean rations (U.K. ZOFRAN tablet over-encapsulated/U.S. ZOFRAN tablet) of the area under the plasma concentration vs. time curve (AUC) from zero to infinity and maximum plasma concentration (Cmax) for ondansetron each lie within the interval 0.80 to 1.25; Geometric Mean Ratio = 0.991, 95% CI 2-sided [0.873 to 1.126] — Geometric Mean Ratio (Treatment OE U.K. tablet / Treatment U.S. tablet)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ondansetron
Time Frame: 24 hours post dose
Population: All study participants (N=12)
Measure: Least Squares Mean (Standard Deviation); unit: nM
Arm/Group | Treatment OE U.K. Tablet | Treatment U.K. Tablet | Treatment U.S. Tablet
Number analyzed (Participants) | 12 | 12 | 12
nM | 82 (18) | 93 (16) | 86 (20)
Statistical Analysis 1: Comparison: Treatment OE U.K. Tablet vs Treatment U.K. Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Study Secondary Hypothesis: A single dose of U.K. ZOFRAN (ondansetron) 8-mg table over-encapsulated is bioequivalent to a single dose of the U.K. ZOFRAN (ondansetron) 8-mg tablet. That is, the true geometric mean ratios (U.K.) ZOFRAN tablet over-encapsulated/U.K. ZOFRAN tablet) of the area under the plasma concentration vs. time curve (AUC) from zero to infinity and maximum plasma concentration (Cmax) for ondansetron each lie within the interval 0.80 to 1.25; Geometric Mean Ratio = 0.886, 95% CI 2-sided [0.813 to 0.966] — Geometric Mean Ratio (Treatment OE U.K. tablet / Treatment U.K. tablet)
Statistical Analysis 2: Comparison: Treatment OE U.K. Tablet vs Treatment U.S. Tablet; Treatment OE U.K. tablet: an over-encapsulated single 8-mg tablet of United Kingdom (U.K.) ZOFRAN (ondansetron) taken orally. Treatment U.S. tablet: a single 8-mg tablet of ZOFRAN (ondansetron) which is marketed in the United States (U.S.) taken orally; Test type: Non-Inferiority or Equivalence — § Study Primary Hypothesis: A single dose of the U.K. ZOFRAN (ondansetron) 8-mg tablet over-encapsulated is bioequivalent to a single dose of the U.S. ZOFRAN (ondansetron) 8-mg tablet. That is, the true geometric mean rations (U.K. ZOFRAN tablet over-encapsulated/U.S. ZOFRAN tablet) of the area under the plasma concentration vs. time curve (AUC) from zero to infinity and maximum plasma concentration (Cmax) for ondansetron each lie within the interval 0.80 to 1.25; Geometric Mean Ratio = 0.951, 95% CI 2-sided [0.872 to 1.037] — Geometric Mean Ratio (Treatment OE U.K. tablet / Treatment U.S. tablet)

ADVERSE EVENTS:
Time Frame: Treatment Period 1, Day 1 to 14 days Post Last Dose of Study Drug in Treatment Period 3, including the 7 day washout in between periods.
Arm/Group | Treatment OE U.K. Tablet | Treatment U.K. Tablet | Treatment U.S. Tablet
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment OE U.K. Tablet (N=12) | Treatment U.K. Tablet (N=12) | Treatment U.S. Tablet (N=12)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.